CLINICAL TRIAL: NCT05232513
Title: The Effect of Hand Massage Applied Before Cataract Surgery on Anxiety, Surgical Fear, Pain and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yağmur Sezer Efe, Assist. Prof. Yağmur Sezer Efe, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/500
Record Dates: First submitted 2021-12-24; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cataract Surgery
Keywords: Anxiety; Fear of surgery; Pain; Hand massage; Cataract surgery
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Hand massage
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand massage group (Experimental): The group that received hand massage for 10 minutes before cataract surgery
  Interventions: Other: Hand massage
- Control group (No Intervention): standard care group

INTERVENTIONS:
Other: Hand massage — Hand massage is an initiative that improves the communication between the massager and the individual, reduces anxiety, and provides comfort and relaxation.
  Arms: Hand massage group

SUMMARY:
ABSTRACT Objective: The research was conducted as a prospective randomized controlled experimental study to determine the effect of hand massage applied before cataract surgery on anxiety, surgical fear, pain and physiological parameters of patients.

Study design: The sample of the study consisted of 60 patients, 30 experimental and 30 control, who had cataract surgery and met the study criteria in Eye Operating Room of a tertiary hospital between 24 December 2020 and 31 May 2021. Ethics committee, institutional permission and participant consent were obtained in this study, and data were collected using the descriptive characteristics form, Physiological Parameters Observation Form (PPOF), VAS-Anxiety, Surgical Fear Scale (SFS), and VAS-Pain scale. In the study, individuals in the experimental group were given hand massage for 10 minutes before cataract surgery. Before and after hand massage, PPOF, VAS-Anxiety and SFS were measured and recorded. In addition, PPOF, VAS-Anxiety and VAS-Pain were measured and recorded again at the postoperative 30th minute. Pearson chi-square, Shapiro Wilk, Levene test, Two-Way Analysis of Variance in Repeated Measurements, Mann-Whitney U test were used in the analysis of the data.

DETAILED DESCRIPTION:
This prospective randomized controlled experimental study is planned in order to determine the effect of hand massage applied before cataract surgery on patients' anxiety and fear of surgery, pain and physiological parameters.

The sample of the study consisted of 60 patients, 30 experimental and 30 control, who had cataract surgery and met the study criteria in Eye Operating Room of a tertiary hospital between 24 December 2020 and 31 May 2021. Ethics committee, institutional permission and participant consent were obtained in this study, and data were collected using the descriptive characteristics form, Physiological Parameters Observation Form (PPOF), VAS-Anxiety, Surgical Fear Scale (SFS), and VAS-Pain scale. In the study, individuals in the experimental group were given hand massage for 10 minutes before cataract surgery. Before and after hand massage, PPOF, VAS-Anxiety and SFS were measured and recorded. In addition, PPOF, VAS-Anxiety and VAS-Pain were measured and recorded again at the postoperative 30th minute. Pearson chi-square, Shapiro Wilk, Levene test, Two-Way Analysis of Variance in Repeated Measurements, Mann-Whitney U test were used in the analysis of the data.

The mean VAS-Anxiety score of the individuals in the experimental group after hand massage was 1.56±1.07, while the control group was 2.80±2.21 (p<0.05); While the VAS-Pain score of the experimental group was 1.00 (2.00), it was 2.00 (1.00) for the control group (p<0.05). It was determined that the mean total score of SFS of the individuals in the experimental group after hand massage was lower than the scores of the individuals in the control group (p<0.05). It was determined that the respiratory and systolic blood pressure values of the patients in the experimental group decreased after hand massage compared to the control group (p<0.05). It was determined that the pulse, SPO2, diastolic blood pressure (DBP) values of the patients in the experimental group after hand massage were not statistically significant compared to the control group (p>0.05). However, it was determined that the pulse and DBP values of the experimental group decreased after the hand massage compared to the values before the hand massage, while the SPO2 value increased.

According to these results; It was determined that hand massage applied before the surgery reduced the patients' anxiety and fear of surgery, positively affected their physiological parameters and reduced the pain levels of the patients. It may be recommended to apply hand massage before surgery in cataract and other surgeries to be performed under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* The 18-80 years old,
* Cataract surgery will be performed using local anesthesia,
* Collaborative and without communication problems (language problems, speech and hearing problems, etc.),
* Those who are conscious and able to answer questions and do not have any disorder/disease (dementia, Alzheimer's, psychological disorder, etc.)
* Open wounds on the skin or those who do not have an obstacle to massage (edema, abscess, skin infection with necrosis, thrombophlebitis, occlusive artery disease, loss of sensation in the hand, neuropathy, mass, fracture and ingrown nails, etc.),
* Does not have psychiatric diseases such as anxiety disorder, panic attack, depression,
* Not receiving any psychiatric treatment such as antipsychotic/anxiolytic,
* Type 1 Diabetes patients who do not develop diabetic neuropathy (under 15 years of age, Type 2 Diabetes patients who have not completed 10 years of age),
* Patients who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* <18 and >80 years old,
* who will undergo cataract surgery under general anesthesia,
* Having previously undergone cataract surgery,
* Having communication problems (language problems, speech and hearing problems, etc.),
* Having a history of LVH with advanced paralysis,
* Those who are not conscious, unable to answer questions, have any disorder/disease (dementia, Alzheimer's, psychological disorder, etc.)
* Open wound on the skin or an obstacle to massage (edema, abscess, skin infection with necrosis, thrombophlebitis, occlusive artery disease, loss of sensation in the hand, mass, fracture and ingrown nails, neuropathy, etc.),
* Having psychiatric diseases such as anxiety disorder, panic attack, depression,
* Receiving psychiatric treatment such as antipsychotic/anxiolytic,
* Type 1 Diabetes patients who have developed diabetic neuropathy (over 15 years, Type 2 Diabetes patients who have completed 10 years),
* Patients who did not volunteer to participate in the study were not included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Surgical Fear Questionnaire (SFQ) scores | before and immediately after the hand massage
  SFQ is scored between 0-10, and an increase in the score from the scale indicates that the patients' fear of surgery increases.
Visual Analogue Scale (VAS)-Anxiety scores | before and immediately after the hand massage, and postop 30.th minutes
  According to the Visual Analogue Scale (VAS)-Anxiety, a high score indicates a high anxiety.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS)-Pain scores | postop 30.th minutes
  According to the Visual Analogue Scale (VAS)-Pain, a high score indicates a high pain.
Physiological parameters-blood pressure | before and immediately after the hand massage, and postop 30.th minutes
  systolic and diastolic blood pressure
Physiological parameters-respiratory rate | before and immediately after the hand massage, and postop 30.th minutes
  respiratory rate
Physiological parameters-pulse rate | before and immediately after the hand massage, and postop 30.th minutes
  pulse rate
Physiological parameters-oxygen saturation | before and immediately after the hand massage, and postop 30.th minutes
  oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Sezer Efe, Assist. Prof., Principal Investigator — ErciyesUniversity
Locations (1):
- Erciyes university, Kayseri, Turkey (Türkiye)